## Wright Foot & Ankle Post-Market Observational Study Statistical Analysis Plan (SAP)

CLINICAL INVESTIGATION TITLE: Wright Foot & Ankle Post-Market Observational Study

**DEVICE NAME:** 611 Nail

BIOARCH

BIOFOAM Ankle Spacer BIOFOAM Wedge System CHARLOTTE MUC Screws CHARLOTTE Quick Staple CHARLOTTE Snap-Off Screws

CLAW II

**DARCO Headed Rearfoot Screws** 

DARCO Headed Screws DARCO Headless Screws

DARCO MFS DARCO MRS

DARCO Plantar Lapidus Plate

DART-FIRE FUSEFORCE FUTURA CSI G-FORCE

**GRAVITY SYNCHFIX** 

**HV Screws** 

MaxLock Edgelock Plate MiniMaxLock ISO Plate

MICA Screws

NEXFIX Snap-Off Screws Omni Evolution Screws ORTHOLOC 2 Ankle Fracture ORTHOLOC 2 CROSSCHECK ORTHOLOC 2 Small Bones ORTHOLOC 3Di Ankle Fusion ORTHOLOC 3Di Hallux

ORTHOLOC 3Di Midfoot/Flatfoot ORTHOLOC Forefoot Fracture ORTHOLOC Plantar Lapidus ORTHOLOC Calc Fracture

PHALINX PITON PRO-TOE VO SALVATION ExFix

SALVATION Bolts and Beams SALVATION 3Di Plates

**SWANSON Toes** 

Telya

UNIMA EVO and NEUTRA Screws

VALOR Nail

STATISTICAL ANALYSIS PLAN

(SAP) VERSION:

1

CLINICAL INVESTIGATION PLAN

(CIP) VERSION:

Z

ClinicalTrials.Gov NCT04118894

**INDICATIONS:** 

The Instructions for Use (IFU) for each individual product can be found at http://www.wright.com/prescribing-use-3.

CLINICAL INVESTIGATION

**DESIGN:** 

Post-Market,

• Multicenter,

• Prospective,

• Non-Randomized

**CONFIDENTIALITY STATEMENT:** 

This Statistical Analysis Plan contains confidential information and its' use is limited to investigational staff intending to conduct the clinical investigation, Institutional Review Boards (IRBs)/Ethics Committees (ECs) and any others charged with reviewing the clinical investigation.

**DATE:** 07-Dec-2021

## **Approval Page**

| Name | Signature | Date | |
|---|---|---|---|
| Jennifer Seidman | Signing Reason: I approve this | document | 45 AM PST |
| Jovi Quiton | Signing Time: 12-Jan-2022 6: 图5记录设施设施设施。 Mg.utm Signer Name: Jovi Quiton Signing Reason: I approve this | 45 AM PST<br>7EFBE9D74<br>12-Jan-2022 9<br>document | :16 AM PST |
| Rebecca Gibson | 74CDF10AA94943E682E55B8 DocuSigned by: Retecte Gibson Signer Name: Rebecca Gibson Signing Reason: I approve this | 384F9F9F96<br>12-Jan-2022 1 | .2:30 PM ES |
| | Jennifer Seidman Jovi Quiton | Jennifer Seidman DocuSigned by: Jentifer Seidman Signer Name: Jennifer Seidman Signing Reason: I approve this Signing Time: 12-Jan-2022 6: DocuSigned by: Jentifer Seidman Signing Reason: I approve this Signing Reason: I approve this Signing Time: 12-Jan-2022 9: Rebecca Gibson Rebecca Gibson Signer Name: Rebecca Gibson Signing Reason: I approve this Signing Reason: I approve this | Jennifer Seidman DocuSigned by: 12-Jan-2022 6: Jennifer Seidman Signing Reason: I approve this document Signing Time: 12-Jan-2022 6:45 AM PST Jovi Quiton Signer Name: Jovi Quiton Signing Reason: I approve this document Signing Reason: I approve this document Signing Time: 12-Jan-2022 9:16 AM PST Rebecca Gibson Rebecca Gibson 74CDF10AA94943E682E55B884F9F9F96 DocuSigned by: 12-Jan-2022 1 Reference Gibson |

## **Table of Contents**

| 1. | Admin | istrative Information | 6 |
|---|---|---|---|
| | 1.1. | LIST OF ABBREVIATIONS | 6 |
| | 1.2. | STATISTICAL ANALYSIS PLAN REVISION HISTORY | 6 |
| | 1.3. | ROLES AND RESPONSIBILITIES | 6 |
| 2. | Introd | uction | 7 |
| | 2.1. | BACKGROUND AND RATIONALE | 7 |
| | 2.2. | CLINICAL INVESTIGATION DESIGN | 7 |
| 3. | Statist | ical Procedure | 8 |
| | 3.1. | FRAMEWORK | 8 |
| 4. | Metho | ds | 9 |
| | 4.1. | RANDOMIZATION | 9 |
| | 4.2. | STATISTICAL INTERIM ANALYSES AND STOPPING GUIDANCE | 9 |
| | 4.3. | TIMING OF FINAL ANALYSES | 9 |
| | 4.4. | TIMING OF OUTCOME ASSESSMENT | 9 |
| | 4.5. | STATISTICAL SOFTWARE | 10 |
| | 4.6. | MISSING DATA | 10 |
| | 4.7. | UNITS | 11 |
| | 4.8. | CALCULATIONS AND TRANSFORMATIONS | 11 |
| 5. | Popula | ntion and Progress | 11 |
| 6. | Analys | is | 11 |
| | 6.1. | Patient Accounting | 11 |
| | 6.2. | Baseline Characteristics | 11 |
| | Subj | ect eligibility | 11 |
| | Dem | ographic | 11 |
| | Med | ical Conditions | 11 |
| | 6.3. | Protocol Deviations | 12 |
| | 6.4. | Intra-operative Factors | 12 |
| | 6.5. | Effectiveness | 12 |
| | 6.6. | HARMS AND SAFETY | 13 |
| 7. | Listing | S | 13 |
| 8. | Appen | dices | 14 |
| | 8.1. | Appendix 1. List of Wright medical devices included in the study. | 14 |

| ADJCHT FOOT 0 | ANIZI E DOCT MADIZET | ODCEDUATIONAL | CTUDY CAD Variation 1 |
|---|---|---|---|
| WKIGHI FUUI &. | ANKLE PUST-MAKKET | OBSERVATIONAL | STUDY SAP - Version 1 |

| Page | 5 | of | 30 |
|------|---|----|----|

| | 8.2. | Appendix 2 - Listing of Tables and Listings, Table Templates | 5 |
|---|---|---|---|
| 9. | Refere | nces | 30 |

## 1. Administrative Information

### 1.1. LIST OF ABBREVIATIONS

| <u>Acronym</u> | <u>Definition</u> |
|---|---|
| ADE | Adverse Device Event |
| AE | Adverse Event |
| CI | Confidence Interval |
| CIP | Clinical Investigation Plan |
| CRF | Case Report Form |
| eCRF | Electronic Case Report Form |
| EC | Ethics Committee |
| EDC | Electronic Data Capture |
| EQ-5D | A standardized health-related quality of life instrument by the EuroQuol Group |
| EU MDR | European Medical Device Regulation |
| FAAM | Foot and Ankle Ability Measure |
| FR | Final Report |
| FU | Follow-Up |
| ICF | Informed Consent Form |
| ICH-GCP | International Conference of Harmonisation Good Clinical Practice |
| IFU | Instructions for Use |
| ITT | Intent-to-Treat |
| Intra-Op | Intra-Operative |
| IR | Interim/Annual Report |
| IRB | Institutional Review Board |
| LTFU | Lost to Follow-Up |
| Op | Operative |
| PP | Per Protocol |
| Post-op | Post-Operative |
| Pre-Op | Pre-Operative |
| SADE | Serious Adverse Device Effect |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |

#### 1.2. STATISTICAL ANALYSIS PLAN REVISION HISTORY

Unanticipated Adverse Device Effect

| Version | Effective Date | Description | Reason |
|---------|-----------------|-----------------|--------|
| 1 | 12 January 2022 | Initial Version | n/a |

### 1.3. ROLES AND RESPONSIBILITIES

UADE

| Role | Contributor | Affiliation |
|---|---|---|
| Author/ Clinical Investigation<br>Manager (CIM) | Jennifer Seidman | Stryker |
| (Senior) Statistician | Jovi Quiton | Stryker |
| Clinical Research Head (CRH) | Rebecca Gibson | Stryker |

## 2. Introduction

#### 2.1. BACKGROUND AND RATIONALE

The European Union (EU) Medical Device Regulation (MDR) 2017/83/EC applies to all medical device manufactures who intend to market their products in the EU. The EU MDR has increased the requirements for clinical data needed for products to maintain certification. Under the regulation, the manufacture must proactively collect and evaluate clinical data to establish and verify:

that under normal conditions of use, a device achieves the performance intended as specified by the manufacturer:

- the clinical benefits of a device as specified by the manufacturer;
- the clinical safety of the device;
  - o Identify previously unknown side-effects;
  - Monitor the intended side-effects and contraindications;
  - o Identify and analyze emerging risks on the basis of factual evidence;
- ensure the continued acceptability of the benefit / risk ratio; and
- systemic misuse or off-label use with a view to verify the intended purpose is correct.

Wright Medical is conducting this observational study to meet the clinical data requirements for the EU MDR.

The purpose of this post-market clinical observational study is to demonstrate the safety and performance of the Wright product after implantation over a standard follow-up period using patient reported outcome measures (PROMs) related to quality of life and functional improvements, safety of the implants, as well as radiographic assessments (X-Rays).

The outcome measures collected in this study will be analyzed and reported as required for local, regional, and country requirements (i.e., regulatory authorities and notified bodies).

#### 2.2. CLINICAL INVESTIGATION DESIGN

This investigation is a global, multi-center, post-market observational study. The study planned to enroll 40 patients per device according to sample size calculations based on the EQ-5D (See study protocol). The enrollment period is expected to be 5 years. Based on the varied definitions of clinical lifetime for each device, the follow-up (FU) period will range 12 weeks to 10 years.

Data will be collected at baseline, surgery, at last scheduled standard of care and/or surgeon release FU time point. Additionally, PROMs and safety may be followed yearly to sufficiently assess the safety of the product over the clinical lifetime as needed based on the current risk analysis for the product.

#### 3. Statistical Procedure

#### 3.1. FRAMEWORK

The purpose of this statistical analysis plan is to guide the analysis and production of statistical output for the Wright Foot & Ankle Post-Market Observational Study. The company decided to discontinue enrollment to the study on November 1, 2021. At study end date, there were 122 patients enrolled in the study. The sample size of 40 patients per device that was originally planned in the study was therefore not met.

The study required at least 40 sample size for each Wright medical device (See INT19-MDR-001 Protocol. Version 3). For the same sample size parameters in the protocol n=10, will yield a power of 0.5. Thus, for the purpose of reporting statistically valid outcomes, descriptive summary statistics will be presented for Wright devices implanted in at least 10 patients enrolled in the study. Patient data on devices that has less than 10 implanted patients will be provided in the listings to be made available for future study or reference. Appendix Table 1 lists the Wright devices that are included in the study.

As the goal of the study is to determine the performance and safety of each device under investigation, analysis of outcomes will be done for each device the patient received. Note that a patient may have received more than one of the Wright devices. In all analysis of outcomes, patient level data will be included in the analysis for each device he/she received.

All analysis to be conducted are of descriptive nature only. No test of hypothesis will be performed. All quantitative variables, including those based on calculations (i.e., improvement from baseline), will be analyzed with a case summary evaluation before the detailed characteristics and parameter can be evaluated. A case summary contains a listing of the number of valid cases/values, missing cases/values (if any) and total cases/values in the specific analysis. The mean and median will be reported to assess the average or centrality of quantitative variables. Improvement from baseline in patient reported outcome (PROM) will be assessed at each post-surgery visit. Improvement will be based on the difference in raw scores.

Whenever the available data allows, the standard deviation, interquartile range (IQR) and maximum and minimum will be calculated. All quantitative variables will be assessed for normality via the Shapiro-Wilk test. The 95% confidence interval (CI) of the mean will be presented when the normality of the data is met.

All qualitative variables, including those based on summaries (secondary elements), will be analyzed listing the proportions, frequencies, column and row totals and missing proportion (if any).

The proportion of device surviving at each visit will be summarized for each device. Rates will be computed based on available data. Missing data will not be imputed.

No imputations for missing data will be conducted.

#### 3.1.1. Primary Analysis / Endpoint

Improvements in subject quality of life after surgery will be assessed by constructing 95% confidence interval for the mean change from baseline score in EQ-5D-5L.

#### 3.1.2. Secondary Analyses

FAAM score improvements from baseline will be summarized with 95% confidence interval for the mean.

Safety of Wright medical products will be assessed by the frequency and rates of the with collected AE safety profiles.

Surgeon and patient assessment of Wright devises will be presented descriptively.

#### 3.1.3. Additional Analyses

Additional Analyses are outlined in the subsequent sections. Analysis details (variables, level of measurement, planned steps) are listed in-depth in the SAP.

- Fusion/Consolidation time for applicable devices
- Deformity Correction for applicable devices

#### 4. Methods

#### 4.1. RANDOMIZATION

No randomization was implemented in the study. A consecutive series of subjects at each site meeting all the eligibility criteria will be enrolled in this clinical investigation.

#### 4.2. STATISTICAL INTERIM ANALYSES AND STOPPING GUIDANCE

Interim analyses will be performed on an annual basis. The progress of the clinical investigation will be reported together with the interim results on the variable level according to the analysis plan.

There will be no stopping rules specified for this clinical investigation.

#### 4.3. TIMING OF FINAL ANALYSES

The full final report with complete analyses, progress and conduct reporting will be created at the end of this clinical investigation.

#### 4.4. TIMING OF OUTCOME ASSESSMENT

Data will be collected at baseline, surgery, at last scheduled standard of care and/or surgeon release FU time point. Additionally, PROMs and safety may be followed yearly to sufficiently assess the product over the clinical lifetime as needed based on the current risk analysis for the product.

The follow-up evaluations will include assessment of device-related adverse events/incidents, evaluation per EQ-5D-5L and FAAM scores as well as surgeon surveys. See the section below for visit windows and a list of assessments to be performed at each visit, given by the CIP.

Table 4.4.1: Assessments and Clinical Investigation Elements

| Procedures | Pre-op/ | Final Clinical | 1-10 yr | Study |
|---|---|---|---|---|
| | Op | Follow-Up | (-/+1 yr) | Close |
| | | Visit | (yearly as | |
| | | (Op to 1yr) | necessary) <sup>4</sup> | |
| Informed Consent | X | | | |
| Inclusion/Exclusion Criteria | X | | | |
| Medical | X | | | |
| History/Demographics | | | | |
| Operative (Surgical) | X | | | |
| procedure/device | | | | |
| EQ-5D | X | X | X | |
| FAAM | X | X | X | |
| Surgeon Survey with | | X | | |
| radiographic assessment | | 11 | | |
| Adverse Event Assessment | X | X | X <sup>3</sup> | |
| Patient Survey | | | X | |
| End of Study | | | | X |
| Surgical Intervention <sup>1</sup> | | | | |
| *Sponsor-approved | | | | |
| Unscheduled Visit <sup>2</sup> | | | | |

<sup>1&</sup>amp;2 These are not scheduled time point events but will be observed throughout study participation

#### 4.5. STATISTICAL SOFTWARE

All statistical analyses will be performed using SAS Version 9.4 or higher on a SAS PC platform.

#### 4.6. MISSING DATA

The intent is to collect as complete a dataset as possible. Nevertheless, in some situations missing data cannot be avoided. The reports and tables therefore will show the number and percentage of missing cases for each analyzed variable in relation to the enrolled cases for each post-operative assessment.

Missing data will be reported for each variable or calculation (if any) and overall totals will be reported including the proportion of missing data (if any).

<sup>&</sup>lt;sup>3</sup> Only required when patient survey indicates an adverse event occurred

<sup>&</sup>lt;sup>4</sup> Follow-up time points only executed if needed per device clinical lifetime definition

#### **4.7.** UNITS

See analysis chapter for details related to units used for the different variables and calculations. In case of collection of variables with non-SI units (i.e., pounds instead to kilograms), conversion of such data into SI units (and vice versa) will be ensured and both results will be reported for the full set of available subjects next to each other in the interim/annual and/or final reports.

#### 4.8. CALCULATIONS AND TRANSFORMATIONS

Distances between times and differences between score results will be calculated. For full details of variables used for calculations and the creation of new variables based on these calculations, see analysis chapter.

## 5. Population and Progress

All analysis will include all subjects implanted with any of the Wright devices listed in Appendix 1, hence called Treated population.

## 6. Analysis

This section will contain the instructions for data analysis and table templates of the presentation of statistical analysis results. The components of the table template will guide the statistical programming and report generation.

#### 6.1. Patient Accounting

See <u>Table 1.1</u>. A summary of subject disposition will be made, noting the number who attended the baseline visit, had the surgery visit by Wright device implanted/used, and then subsequently attended the remaining study visits.

#### 6.2. Baseline Characteristics

#### Subject eligibility

See <u>Table 1.2</u>. The inclusion and exclusion criteria will be summarized for the treated population in order to assess adherence or deviation of subjects to the study eligibility.

#### **Demographic**

See <u>Table 1.3</u>. Demographics and clinical characteristics at baseline will be summarized descriptively, and will include the following: Age, Race; Gender; Height in cm; Weight in kg, BMI  $(kg/m^2)$  and smoking status. Age in years will be calculated as:

age = FLOOR((INTCK('month',BRTHDT,INFCONDT) - (day(INFCONDT) < day(BRTHDT))) / 12);

#### **Medical Conditions**

See <u>Table 1.4</u>. The pre-operative relevant medical conditions will be summarized by frequency and proportion for each Wright device.

#### 6.3. Protocol Deviations

See Table 1.5. Deviations from the protocol that occurred during the conduct recorded for each patient will be summarized by frequency and rate of occurrence.

#### 6.4. Intra-operative Factors

See <u>Table 2.1</u>. The operative information will be summarized descriptively and will include the following: indication for use, prior surgery, location of surgery.

#### 6.5. Effectiveness

#### 6.5.1. Primary endpoint analysis: EQ-5D

See <u>Table 3.1</u>. EQ-5D is the primary endpoint of the study. EQ-5D is generic health survey that can be used to compare improvement across different interventions—and measure changes in health-related quality of life over time. Three language versions of the EQ-5D questionnaire: English, German and France were used. The scores regardless of language will be combined in the analysis. The EQQ-5D Two components of the EQ-5D will be summarized: Index value and overall health score. The five (5) health state measure in the EQ-5D questionnaire will be used to calculate the EQ-5D index value. An EQ-5D for patient standardized for the country origin will be computed based on the total score of the health measures. The country-specific EQ-5D reference scores will be obtained from EuroQoL Group (<a href="www.euroqol.org">www.euroqol.org</a>). A high EQ-5D index value indicates a better health state while a low EQ-5D index value indicates a wore health state. On the other hand, the Eq-5D overall health score, ranges from 0 to 100, is a single measure of the patient's assessment of their current health status. Higher score indicates better health state while a low score indicates a worse health state.

#### 6.6.2 Secondary endpoints

#### **FAAMS**

See <u>Table 3.2.1</u> The Foot and Ankle Ability Measure (FAAM) is a self-report outcome instrument to assess physical function for individuals with foot and ankle related impairments. Like the EQ-5D, three language versions of the FAAM questionnaire were used. The FAAM consists of 29-item questions divided into two subscales: 21-item activities of daily living (ADL) subscale, 8-item sports subscale. Each item is scored on a 5-point Likert scale (4 to 0) from 'no difficulty at all' to 'unable to do'. Responses of "not applicable" are not counted. The score on each of the items are added together to get the subscale total score. The ADL subscale total score range from 0 to 84 and 0 to 32 for the sports subscale. The patient score for the ADL and sports subscale will be transformed to percentage scores by considering the highest possible score for non-missing items. Higher score indicates hinger level of function for each subscale, with 100% representing no dysfunction (Martin et al., 2009).

See <u>Table 3.2.2</u> Patients assessed their current level of function as Normal, Nearly Normal, Abnormal, or Severely Abnormal. Summaries will be presented for each Wright device and visit.

#### SURGEON ASSESSMENT AND RADIOGRAPHIC OUTCOME

See <u>Table 4.1</u>. At the final visit of the patient, the attending surgeon assessed the surgical foot to assess the outcome. The surgeon also assessed the radiographic outcome of the surgery. For each Wright device of interest, the following will be summarized:

- Days from surgery to radiographic evaluation
- Imaging procedure done: standing AP/lateral, hindfoot alignment view, CT, MRI, Other
- Surgeon opinion on Wright product performance
- Bony union outcome for joint arthrodesis device

See <u>Table 4.2</u>. The surgeon assessment of angle deformity correction based on radiograph will be summarized for the following:

- Angle deformity correction for hallux valgus deformity: Halux Valgus angle, Intermetatarsal angle, Distal Metatarsal Articular Angle
- Angle deformity correction for flatfoot or charcot: Mearys angle, Talonavicular Angle, Other
- Surgeon observed adverse event (Y/N)

#### 6.6. HARMS AND SAFETY

See <u>Table 5.1</u>. The safety of each device will be summarized in the interim and final report. Overall summary of adverse events will be presented for each device. Total frequencies and percentages of adverse events for each Wright device will be summarized for the following factors:

- i.) Procedure-Related Adverse Event / Incident.
- ii.) Device-Related Adverse Event / Incident
- iii.) Device Failure
- iv.) Unanticipated Adverse Device Event
- v.) Serious Adverse Event (SAE)
- vi.) Hospitalization SAE Outcome
- vii.) Treatment Required for the AE

The occurrence and rate of SAE will be further categorized by the outcome of the SAE (i.e., death, hospitalization).

The rates for device failure will be the basis of the survival rates for each device. The above AE factors will also be summarized for each study site.

#### 7. Listings

Appendix II contains the contents of Listing of Tables (Appendix 2A), Listings (Appendix 2C and Figures (Appendix 2D). All patient data listings will include page-breaks at the beginning of each investigative site to allow simple partitioning of the listing data by site.

All listings will contain the following standard elements: study name and protocol number, title of display, data version date, and data analysis date.

## 8. Appendices

8.1. Appendix 1. List of Wright medical devices included in the study.

| | Fall and the Time a Bank at |
|-------------------------------|---------------------------------|
| Device C11 Net | Follow-Up Time Period |
| 611 Nail | 1 year |
| BIOARCH | 1 year, 2 year |
| BIOFOAM Ankle Spacers | 1 year |
| BIOFOAM Wedge System | 1 year |
| CHARLOTTE MUC Screws | 1 year |
| CHARLOTTE Quick Staple | 1 year |
| CHARLOTTE Snap-Off Screws | 1 year |
| CLAW II | 1 year |
| DARCO Headed Screws | 1 year |
| DARCO Headless Screws | 1 year |
| DARCO MFS | 1 year |
| DARCO MRS | 1 year |
| DARCO Plantar Lapidus Plate | 1 year |
| DART-FIRE | 1 year |
| FUSEFORCE | 1 year |
| FUTURA CSI | 1 year, 2 year |
| G-FORCE | 1 year, 2 year |
| GRAVITY SYNCHFIX | 1 year, 2 year |
| HV Screws | 1 year |
| MaxLock Edgelock Plate | 1 year |
| MiniMaxLock ISO Plate | 1 year |
| MICA Screws | 1 year |
| NEXFIX Snap-Off Screws | 1 year |
| Omni Evolution Screws | 1 year |
| ORTHOLOC 2 Ankle Fracture | 1 year |
| ORTHOLOC 2 CROSSCHECK | 1 year |
| ORTHOLOC 2 Small Bones | 1 year |
| ORTHOLOC 3Di Ankle Fusion | 1 year |
| ORTHOLOC 3Di Hallux | 1 year |
| ORTHOLOC 3Di Midfoot/Flatfoot | 1 year |
| ORTHOLOC Forefoot Fracture | 1 year |
| ORTHOLOC Plantar Lapidus | 1 year |
| ORTHOLOC Calc Fracture | 1 year |
| PHALINX | 1 year |
| PITON | 1 year |
| PRO-TOE VO | 1 year |
| SALVATION ExFix | 1 year |
| SALVATION Bolts and Beams | 1 year |
| SALVATION 3Di Plates | 1 year |
| SWANSON Toes | 1 year, 2 year, 3 year, 4 year, |
| | 5 year, 6 year, 7 year, 8 year, |
| | 9 year, 10 year |
| Telya | 1 year |
| UNIMA EVO and NEUTRA Screws | 1 year |
| VALOR Nail | 1 year |
| · | ) |

## 8.2. Appendix 2 - Listing of Tables and Listings, Table Templates

### A. LISTING OF TABLES

| Table | 1.1 | Subject Accounting |
|---|---|---|
| Table | 1.2 | Subject Eligibility |
| Table | 1.3 | Demographics and Clinical Characteristics |
| Table | 1.4 | All Protocol Deviations |
| Table | 1.5 | Medical History |
| Table | 2.1 | Surgical and Operative Information |
| Table | 2.2 | Additional Surgical Procedures Performed |
| Table | 3.1 | EQ-5D by device and visit |
| Table | 3.2.1 | FAAM score by device and visit |
| Table | 3.2.2 | FAAM overall rating by Device and Visit |
| Table | 4.1 | Surgeon assessment by device |
| Table | 4.2 | Radiographic assessment by device |
| Table | 5.1 | Life table for time to first device related adverse event by device |
| Table | 5.2 | Life table for device failure by device |
| Table | 5.3 | Life table for time to death by device |
| Table | 6.1 | Adverse event by device |

#### **B. ANALYSIS TABLE TEMPLATES**

**Table 1.1. Patient Accounting.** 

| | Site | | |
|---|---|---|---|
| | | Post Op Visit Post Op Vis | |
| | Baseline | 1 | 2 |
| Device 1 | | | |
| Total | XX | XX | XX |
| Completers | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Reason for discontinu | ation | | |
| Lost to follow-up | XX | XX | XX |
| Withdrew consent | XX | XX | XX |
| Adverse event | XX | XX | XX |
| Other | XX | XX | XX |
| : | : | : | : |
| Device k | | | |
| Total | XX | XX | XX |
| Completers | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Reason for discontinu | ation | | |
| Lost to follow-up | XX | XX | XX |
| Withdrew consent | XX | XX | XX |
| Adverse event | XX | XX | XX |
| Other | XX | XX | XX |

**Table 1.2. Subject Eligibility** 

| | Inclu | sion Quies | tions | Excl | usion Ques | stins | Eligible |
|---|---|---|---|---|---|---|---|
| | 1 | 2 | 3 | 1 | 2 | 3 | |
| | f(%) | f(%) | f(%) | f(%) | f(%) | f(%) | f(%) |
| All | | | | | | | |
| Sites | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) |
| Site | | | | | | | |
| 1 | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) |
| 2 | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) |
| 3 | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) |
| 4 | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) |
| Total | | | | | | | XX |

 Table 1.3. Demographics and Clinical Characteristics

| Factors | | | | | Freq ( | %) | |
|---|---|---|---|---|---|---|---|
| Gender | | | | | | | |
| Male | | | | | xx(xx.x | (%) | |
| Female | | | | | xx(xx.x | (%) | |
| Smoking | | | | | | | |
| Never | xx(xx.x%) | | | | | | |
| Previous | | | | | | | |
| Current, ≤1 pack/day | | | | | xx(xx.x | (%) | |
| Current, >1 pack/day | | | | | | | |
| | n | mean | sd | min | max | median (IQR) | 95% CI |
| Age (years) | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x(xx.x, xx.x) | (xx.x, xx.x) |
| Weight (kg) | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x(xx.x, xx.x) | (xx.x, xx.x) |
| Height (cm) | XX.X XX.X XX.X XX.X XX.X XX.X(XX.X, XX.X) (XX. | | | | | | (xx.x, xx.x) |
| BMI (kg/m2) | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x(xx.x, xx.x) | (xx.x, xx.x) |

Table 1.4. Medical History

| Factors | Freq (%) |
|------------------------------|-----------|
| Autoimmune Disorder | |
| Cardiovascular Disorder | xx(xx.x%) |
| Respiratory Disorder Skin | xx(xx.x%) |
| Gastrointestinal Disorder | |
| Genitourinary Disorder | xx(xx.x%) |
| Hematological Disorder | xx(xx.x%) |
| Psychological Disorder | xx(xx.x%) |
| Musculoskeletal Disorder | xx(xx.x%) |
| Neurological Disorder | xx(xx.x%) |
| Endocrine/Metabolic Disorder | xx(xx.x%) |
| Subcutaneous Tissue Disorder | xx(xx.x%) |
| Peripheral Vascular Disease | xx(xx.x%) |
| Diabetes | xx(xx.x%) |
| Type I | xx(xx.x%) |
| Type II | xx(xx.x%) |
| Other | xx(xx.x%) |

**Table 1.5. All Protocol Deviations** 

| Type of Deviation | | | | | |
|---|---|---|---|---|---|
| Subjects | Dev 1 | Dev 2 | Dev 3 | Dev 4 | Deviations |
| | Freq (%) | Freq (%) | Freq (%) | Freq (%) | |
| All Subjects (N=xx) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | XX |
| | | | i | i | |
| Wright Device | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | XX |
| Device 1 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | XX |
| Device 1 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | XX |
| : | | | | | |
| Device k | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | XX |

#### Note:

Dev 1 -Visit completed but outside of window

Dev 2-Completely missed follow up visit

Dev 3 -Patient questionnaire(s) not done

Dev 4-Other deviations

**Table 2.1. Surgical and Operative Information** 

| Factors | Device 1 | Device 2 | Device k |
|---------------------------------------|-----------|-----------|-----------|
| | Freq (%) | Freq (%) | Freq (%) |
| Indication for use | | | |
| Post traumatic | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Arthritis | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Fracture | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Fusion | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Reconstruction/Correction | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Revision procedure | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Instability | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Skeletal defect after tumor selection | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Prior surgery | | | |
| Yes | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| No | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Location of Surgery | | | |
| Right | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Left | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |

Table 3.1 EQ-5D by device and visit

| | | Visit | Visit |
|---|---|---|---|
| Wright Device | Baseline<br>(n=xx) | Post-op Visit 1 (n=xx) | Post-op Visit 2<br>(n=xx) |
| Device 1 | | | |
| Overall Health | | | |
| mean±sd | xx.x±xx.x | xx.x±xx.x | xx.x±xx.x |
| median | XX.X | XX.X | XX.X |
| min,max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Index Value | XX.X | XX.X | XX.X |
| mean±sd | xx.x±xx.x | xx.x±xx.x | xx.x±xx.x |
| median | XX.X | XX.X | XX.X |
| min,max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Change from Baseline | | | |
| Overall Health | | | |
| mean±sd | | xx.x±xx.x | xx.x±xx.x |
| median | | XX.X | XX.X |
| min,max | | XX.X, XX.X | XX.X, XX.X |
| 95% CI | | (xx.x, xx.x) | (xx.x, xx.x) |
| Index Value | | XX.X | XX.X |
| mean±sd | | xx.x±xx.x | xx.x±xx.x |
| median | | XX.X | XX.X |
| min,max | | XX.X, XX.X | XX.X, XX.X |
| 95% CI | | (xx.x, xx.x) | (xx.x, xx.x) |
| Device 2 | | , , | |
| Overall Health | | | |
| mean±sd | xx.x±xx.x | xx.x±xx.x | xx.x±xx.x |
| median | XX.X | XX.X | XX.X |
| min,max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Index Value | XX.X | XX.X | XX.X |
| mean±sd | xx.x±xx.x | xx.x±xx.x | xx.x±xx.x |
| median | XX.X | XX.X | XX.X |
| min,max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Change from Baseline | | | |
| Overall Health | | | |
| mean±sd | | xx.x±xx.x | xx.x±xx.x |
| median | | XX.X | XX.X |
| min,max | | XX.X, XX.X | XX.X, XX.X |
| 95% CI | | (xx.x, xx.x) | (xx.x, xx.x) |
| Index Value | | XX.X | XX.X |
| mean±sd | | xx.x±xx.x | xx.x±xx.x |
| median | | XX.X | XX.X |
| min,max | | XX.X, XX.X | XX.X, XX.X |
| 95% CI | | (xx.x, xx.x) | (xx.x, xx.x) |
| , | | (2012) 2012 | (20012) (20012) |

| Device k | | | |
|----------------------|--------------|--------------|--------------|
| Overall Health | | | |
| mean±sd | xx.x±xx.x | xx.x±xx.x | xx.x±xx.x |
| median | XX.X | XX.X | XX.X |
| min,max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Index Value | XX.X | XX.X | XX.X |
| mean±sd | xx.x±xx.x | xx.x±xx.x | xx.x±xx.x |
| median | XX.X | XX.X | XX.X |
| min,max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Change from Baseline | | | |
| Overall Health | | | |
| mean±sd | | xx.x±xx.x | xx.x±xx.x |
| median | | XX.X | XX.X |
| min,max | | XX.X, XX.X | XX.X, XX.X |
| 95% CI | | (xx.x, xx.x) | (xx.x, xx.x) |
| Index Value | | XX.X | XX.X |
| mean±sd | | xx.x±xx.x | xx.x±xx.x |
| median | | XX.X | XX.X |
| min,max | | XX.X, XX.X | XX.X, XX.X |
| 95% CI | | (xx.x, xx.x) | (xx.x, xx.x) |

Table 3.2.1 FAAM score by device and visit.

| Wright device | Base | eline | | | Fol | low-up Vis | it | | Fina | ıl Visit | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | n | mean±sd | min,max | 95% CI | n | mean±sd | min,max | 95% CI | n | mean±sd | min,max | 95% CI |
| Device 1 | | • | | | | | | | • | | | |
| FAAM SANE | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) |
| Sports Subscale | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) | xx | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) |
| ADL Subscale | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) | xx | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) |
| Change from B | aselii | пе | | | | | | | | | | |
| FAAM SANE | | | | | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) |
| Sports Subscale | | | | | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) |
| ADL Subscale | | | | | xx | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) |
| Device 2 | | | | | | | | | | | | |
| FAAM SANE | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) | xx | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) |
| Sports Subscale | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) | xx | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) |
| ADL Subscale | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) | xx | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) |
| Change from B | aselii | ne | | | | | | | | | | |
| FAAM SANE | | | | | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) |
| Sports Subscale | | | | | xx | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) |
| ADL Subscale | | | | | xx | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) |
| : | | | | | | | | | | | | |
| Device k | | | | | | | | | | | | |
| FAAM SANE | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) |
| Sports Subscale | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) |
| ADL Subscale | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) |
| Change from B | aseli | ne | | | | | | | | | | |
| FAAM SANE | | | | | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) |
| Sports Subscale | | | | | xx | xx.x±xx.x | xx.x, xx.x | (xx.x, xx.x) | XX | xx.x±xx.x | xx.x, xx.x | (xx.x, xx.x) |
| ADL Subscale | | | | | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) | XX | xx.x±xx.x | XX.X, XX.X | (xx.x, xx.x) |

Note:

ADL - activities of daily living

SANE - single assessment numeric evaluation

Tale 3.2.2 FAAM overall rating by device and visit

| Wright device | | Base | eline | |
|---|---|---|---|---|
| | Normal | Nearly Normal | Abnormal | Severely<br>abnormal |
| Device 1 | xx/xx (xx.x%) | xx/xx (xx.x%) | xx/xx (xx.x%) | xx/xx (xx.x%) |
| Device 1 | xx/xx (xx.x%) | xx/xx (xx.x%) | xx/xx (xx.x%) | xx/xx (xx.x%) |
| : | | | | |
| Device k | xx/xx (xx.x%) | xx/xx (xx.x%) | xx/xx (xx.x%) | xx/xx (xx.x%) |
| | | Final | Visit | |
| | Normal | Nearly Normal | Abnormal | Severely<br>abnormal |
| Device 1 | xx/xx (xx.x%) | xx/xx (xx.x%) | xx/xx (xx.x%) | xx/xx (xx.x%) |
| Device 1 | xx/xx (xx.x%) | xx/xx (xx.x%) | xx/xx (xx.x%) | xx/xx (xx.x%) |
| : | | | | |
| Device k | xx/xx (xx.x%) | xx/xx (xx.x%) | xx/xx (xx.x%) | xx/xx(xx.x%) |

Table 4.1 Surgeon evaluation by device

| Wright device | Follow- | up Visit | | Fin | al Visit | |
|---|---|---|---|---|---|---|
| | Factors | N | % | Factors | N | % |
| Device 1 | Bony union | | | Bony union | | |
| | Yes | XX | xx.x% | Yes | XX | xx.x% |
| | No | XX | xx.x% | No | XX | xx.x% |
| | | | | Wright product | performed | l as |
| | | | | intended | | |
| | | | | Yes | XX | xx.x% |
| | | | | No | XX | xx.x% |
| Device 2 | | | | | | |
| | Bony union | | | Bony union | | |
| | Yes | XX | xx.x% | Yes | XX | xx.x% |
| | No | XX | xx.x% | No | XX | xx.x% |
| | | | | Wright product intended | performed | las |
| | | | | Yes | XX | xx.x% |
| | | | | No | XX | xx.x% |
| : | | | | | | |
| Device k | | | | | | |
| | Bony union | | | Bony union | | |
| | Yes | XX | xx.x% | Yes | XX | xx.x% |
| | No | XX | xx.x% | No | XX | xx.x% |
| | No | XX | xx.x% | Other | XX | xx.x% |
| | | | | Wright product | performed | l as |
| | | | | intended | | |
| | | | | Yes | XX | xx.x% |
| | | | | No | XX | xx.x% |

Table 4.2 Surgeon assessment of deformity correction based on radiograph by device.

| Wright d | evice | | | Ba | seline | | | | | F | inal v | /isit | | | | Imp | rovem | ent | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | mean | sd | min | max | 95% CI | n | mean | sd | min | max | 95% CI | n | mean | sd | min | max | 95% CI |
| Device 1 | | | | | | | | | | | | | | | | | | | |
| | Degree of deformity co | rrection | | | | | | | | | | | | | | | | | |
| | Hallux valgus procedure | | | | | | | | | | | | | | | | | | |
| | Hallux valgus | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | xx.x | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) |
| | Intermetatarsal Angle | XX.X | XX.X | XX.X | xx.x | xx.x | (xx.x, xx.x) | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | xx.x | xx.x | XX.X | XX.X | XX.X | (xx.x, xx.x) |
| | DMA Angle | XX.X | XX.X | XX.X | xx.x | xx.x | (xx.x, xx.x) | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | xx.x | xx.x | XX.X | XX.X | XX.X | (xx.x, xx.x) |
| | Flatfoot or charcot proced | dure | | | | | | | | | | | | | | | | | |
| | Mearys Angle | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) |
| | TNV Angle | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | xx.x | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | xx.x | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) |
| | Other | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | XX.X | xx.x | XX.X | XX.X | XX.X | (xx.x, xx.x) |
| Device 2 | | | | | | | | | | | | | | | | | | | |
| | Degree of deformity co | rrection | | | | | | | | | | | | | | | | | |
| | Hallux valgus procedure | | | | | | | | | | | | | | | | | | |
| | Hallux valgus | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) |
| | Intermetatarsal Angle | XX.X | XX.X | XX.X | xx.x | xx.x | (xx.x, xx.x) | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | xx.x | xx.x | XX.X | XX.X | XX.X | (xx.x, xx.x) |
| | DMA Angle | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) |
| | Flatfoot or charcot proced | dure | | | | | | | | | | | | | | | | | |
| | Mearys Angle | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) |
| | TNV Angle | XX.X | XX.X | XX.X | XX.X | xx.x | (xx.x, xx.x) | xx.x | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | XX.X | xx.x | XX.X | XX.X | XX.X | (xx.x, xx.x) |
| | Other | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) |
| : | | | | | | | | | | | | | | | | | | | |
| Device k | | | | | | | | | | | | | | | | | | | |
| | Degree of deformity co | rrection | | | | | | | | | | | | | | | | | |
| | Hallux valgus procedure | | | | | | | | | | | | | | | | | | |
| | Hallux valgus | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) |
| | Intermetatarsal Angle | XX.X | XX.X | XX.X | xx.x | xx.x | (xx.x, xx.x) | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | xx.x | xx.x | XX.X | XX.X | XX.X | (xx.x, xx.x) |
| | DMA Angle | XX.X | XX.X | XX.X | xx.x | xx.x | (xx.x, xx.x) | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | xx.x | xx.x | XX.X | XX.X | XX.X | (xx.x, xx.x) |
| | Flatfoot or charcot proced | dure | | | | | | | | | | | | | | | | | |
| | Mearys Angle | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | xx.x | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) |
| | TNV Angle | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | xx.x | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | xx.x | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) |
| | Other | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) | XX.X | XX.X | XX.X | XX.X | XX.X | (xx.x, xx.x) |

Table 5.1 Adverse Events by device.

| Adverse Events | Device | e 1 | | | Device k | |
|---|---|---|---|---|---|---|
| | Subjects<br>(%) | Events | Subjects<br>(%) | Events | Subjects<br>(%) | Events |
| Procedure-Related | xx (xx.x%) | XX | | | xx (xx.x%) | XX |
| Device-Related | xx (xx.x%) | XX | | | xx (xx.x%) | XX |
| Device Failure | xx (xx.x%) | XX | | | xx (xx.x%) | XX |
| Unanticipated AE | xx (xx.x%) | XX | | | xx (xx.x%) | XX |
| Serious AE | xx (xx.x%) | XX | | | xx (xx.x%) | XX |
| Hospitalization | xx (xx.x%) | XX | | | xx (xx.x%) | XX |
| Death | xx (xx.x%) | XX | | | xx (xx.x%) | XX |
| Required Treatment | xx (xx.x%) | XX | | | xx (xx.x%) | XX |
| Physical Therapy | xx (xx.x%) | XX | | | xx (xx.x%) | XX |
| Medication | xx (xx.x%) | XX | | | xx (xx.x%) | XX |
| Surgery | xx (xx.x%) | XX | | | xx (xx.x%) | xx |
| Other | xx (xx.x%) | XX | | | xx (xx.x%) | XX |

## C. LISTING OF LISTINGS

| Listing | 1 | Demographic Information |
|---|---|---|
| Listing | 2 | Inclusion/Exclusion Criteria |
| Listing | 3 | Protocol Deviations |
| Listing | 4 | Medical History |
| Listing | 5 | Surgical and Operative Information |
| Listing | 6 | EQ-5D Score |
| Listing | 7 | FAAMS Score |
| Listing | 8 | Surgeon assessment and radiographic deformity correction assessment |
| Listing | 9 | Adverse Events |
| Listing | 10 | Study Completion |

## 9. References

Domsic RT, Saltzman CL. Ankle osteoarthritis scale. Foot Ankle Int. 1998; 19:466-471 EQ5D-5L Questionnaire; EQ- $5D^{TM}$  is a trade mark of the EuroQol Research Foundation.

Maher, A, Kilmartin, T. An analysis of Euroqol EQ5D and Manchester Oxford Foot Questionnaire. *Journal of Foot and Ankle Research* 2012; 5; 7

Martin RL, Hutt DM, Wukich DK. Validity of the Foot and Ankle Ability Measure (FAAM) in Diabetes Mellitus. Foot Ankle Int. 2009 Apr;30(4):297-302

Wright Foot & Ankle Post-Market Observational Study INT19-MDR-001 Protocol. Version 31-JUL-2019

## **DocuSign**

#### **Certificate Of Completion**

Envelope Id: C050C43F96714D4F9539ABD01D41FCD6

Subject: Please DocuSign: Foot and Ankle Study\_SAP\_FINAL.docx

Source Envelope:

Document Pages: 30 Signatures: 3
Certificate Pages: 5 Initials: 0

AutoNav: Enabled

Envelopeld Stamping: Disabled

Time Zone: (UTC-08:00) Pacific Time (US & Canada)

Status: Completed

Envelope Originator:
Jennifer Seidman
325 Corporate Drive
New Jersey, NC 07430
jennifer.seidman@stryker.com

IP Address: 73.91.139.149

Sent: 1/12/2022 6:44:47 AM

Viewed: 1/12/2022 6:45:06 AM

Signed: 1/12/2022 6:45:28 AM

#### **Record Tracking**

Status: Original

1/12/2022 6:42:08 AM

Holder: Jennifer Seidman

Jennifer Seidman

jennifer.seidman@stryker.com

Location: DocuSign

**Timestamp** 

#### Signer Events

Jennifer Seidman

jennifer.seidman@stryker.com Manager, Clinical Research

Stryker

Security Level: Email, Account Authentication

(Required)

Signature Adoption: Pre-selected Style

Signature ID:

Signature

0F0D41F7-E3FB-4151-8241-9017EFBE9D74

Using IP Address: 73.91.139.149

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 4/13/2021 8:24:54 AM ID: f716f037-0f6b-48c1-a7a6-a6116e5e35db

Jovi Quiton

jovelyn.quiton@stryker.com

Security Level: Email, Account Authentication

(Required)

Jagrita

Sent: 1/12/2022 6:45:32 AM Viewed: 1/12/2022 8:57:49 AM Signed: 1/12/2022 9:16:33 AM

Signature Adoption: Uploaded Signature Image

Signature ID:

74CDF10A-A949-43E6-82E5-5B884F9F9F96

Using IP Address: 64.136.252.163

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 10/5/2021 5:45:00 PM

ID: c715def7-3ace-4067-b9f7-ba2bbac6f969

Rebecca Gibson rebecca.gibson@stryker.com Director, Clinical Operations Stryker Corporation - Trauma & Extremitites Security Level: Email, Account Authentication (Required)

**Signer Events** 

Rebecco Gibson

**Timestamp** Sent: 1/12/2022 9:16:38 AM Viewed: 1/12/2022 9:30:08 AM Signed: 1/12/2022 9:30:39 AM

Signature Adoption: Pre-selected Style

Signature ID:

**Signature** 

B69B71B0-C1FA-437D-B216-59BFBEB69FE2

Using IP Address: 174.247.29.182

Signed using mobile

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 1/12/2022 6:23:35 AM ID: f3080bb8-db99-4d4c-81a3-f26f7c2a3ae7

| In Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent Certified Delivered Signing Complete Completed | Hashed/Encrypted Security Checked Security Checked Security Checked | 1/12/2022 6:44:47 AM<br>1/12/2022 9:30:08 AM<br>1/12/2022 9:30:39 AM<br>1/12/2022 9:30:39 AM |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disclosure | | |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Stryker Corporation - Trauma & Extremities - Part 11 (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through your DocuSign, Inc. (DocuSign) Express user account. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to these terms and conditions, please confirm your agreement by clicking the 'I agree' button at the bottom of this document.

## **Getting paper copies**

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. For such copies, as long as you are an authorized user of the DocuSign system you will have the ability to download and print any documents we send to you through your DocuSign user account for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

## Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

## Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. To indicate to us that you are changing your mind, you must withdraw your consent using the DocuSign 'Withdraw Consent' form on the signing page of your DocuSign account. This will indicate to us that you have withdrawn your consent to receive required notices and disclosures electronically from us and you will no longer be able to use your DocuSign Express user account to receive required notices and consents electronically from us or to sign electronically documents from us.

#### All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through your DocuSign user account all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

#### **How to contact Stryker Corporation - Trauma & Extremities - Part 11:**

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: rebecca.gibson@stryker.com

# To advise Stryker Corporation - Trauma & Extremities - Part 11 of your new e-mail address

To let us know of a change in your e-mail address where we should send notices and disclosures electronically to you, you must send an email message to us at rebecca.gibson@stryker.com and in the body of such request you must state: your previous e-mail address, your new e-mail address. We do not require any other information from you to change your email address.. In addition, you must notify DocuSign, Inc to arrange for your new email address to be reflected in your DocuSign account by following the process for changing e-mail in DocuSign.

To request paper copies from Stryker Corporation - Trauma & Extremities - Part 11 To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an e-mail to rebecca.gibson@stryker.com and in the body of such request you must state your e-mail address, full name, US Postal address, and telephone number. We will bill you for any fees at that time, if any.

To withdraw your consent with Stryker Corporation - Trauma & Extremities - Part 11 To inform us that you no longer want to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your DocuSign account, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may; ii. send us an e-mail to rebecca.gibson@stryker.com and in the body of such request you must state your e-mail, full name, IS Postal Address, telephone number, and account number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

#### Required hardware and software

| Operating Systems: | Windows2000? or WindowsXP? |
|----------------------------|----------------------------------------------|
| Browsers (for SENDERS): | Internet Explorer 6.0? or above |
| Browsers (for SIGNERS): | Internet Explorer 6.0?, Mozilla FireFox 1.0, |
| | NetScape 7.2 (or above) |
| Email: | Access to a valid email account |
| Screen Resolution: | 800 x 600 minimum |
| Enabled Security Settings: | |
| | •Allow per session cookies |
| | •Users accessing the internet behind a Proxy |
| | Server must enable HTTP 1.1 settings via |
| | proxy connection |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, we will provide you with an email message at the email address we have on file for you at that time providing you with the revised hardware and software requirements, at which time you will

have the right to withdraw your consent.

### Acknowledging your access and consent to receive materials electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please verify that you were able to read this electronic disclosure and that you also were able to print on paper or electronically save this page for your future reference and access or that you were able to e-mail this disclosure and consent to an address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format on the terms and conditions described above, please let us know by clicking the 'I agree' button below.

By checking the 'I Agree' box, I confirm that:

- I can access and read this Electronic CONSENT TO ELECTRONIC RECEIPT OF ELECTRONIC RECORD AND SIGNATURE DISCLOSURES document; and
- I can print on paper the disclosure or save or send the disclosure to a place where I can print it, for future reference and access; and
- Until or unless I notify Stryker Corporation Trauma & Extremities Part 11 as described above, I consent to receive from exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to me by Stryker Corporation Trauma & Extremities Part 11 during the course of my relationship with you.